CLINICAL TRIAL: NCT01495325
Title: Effect of Woodsmoke on Vascular Function in Healthy Firefighters
Brief Title: Effect of Woodsmoke on Vascular Function
Acronym: FIREWOOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Umeå University (Other); NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2011-194-31M; PG/11/27/28842 (Other Grant/Funding Number: BRITISH HEART FOUNDATION)
Record Dates: First submitted 2011-10-11; First posted 2011-12-20 (Estimated); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Vascular Function
Keywords: Firefighter; Woodsmoke; Vascular function; Air Pollution; Endothelial function; Thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Filtered Air Exposure (Sham Comparator): 1 hour exposure to filtered air during intermittent exercise
  Interventions: Procedure: Forearm Vascular Study; Procedure: Badimon Chamber
- Woodsmoke Exposure (Active Comparator): 1 hour exposure to dilute woodsmoke at a concentration of 1000µg/m3 during intermittent exercise
  Interventions: Procedure: Forearm Vascular Study; Procedure: Badimon Chamber

INTERVENTIONS:
Procedure: Forearm Vascular Study — Forearm venous occlusion plethysmography to measure forearm blood flow during intra-arterial infusion of the vasodilators Verapamil (10-100 µg/min), bradykinin (100-1000 pmol/min), sodium nitroprusside (2-8 µg/min) and Acetylcholine (5-20 µg/min).
  Other Names: Other Names:; BK; SNP; ACh
Procedure: Badimon Chamber — Ex-vivo assessment of thrombus formation using the Badimon Chamber

SUMMARY:
Exposure to air pollution is a well established risk factor for the development of heart disease. Firefighters are exposed to excess air pollution in the form of wood smoke during the extinguishing of forest or woodland fires. Heart attacks in on-duty firefighters have been linked to specific duties and in particular fire suppression, but the reasons for this increase in risk are not well understood. Exposure to wood smoke may alter blood vessel function and increase blood clot formation to explain the link between fire suppression and heart attacks.

The investigators wish to determine the effect of exposure to wood smoke at concentrations found at the perimeter of a woodland fire on blood vessel function and clotting in healthy non-smoking male professional firefighters or volunteers. Volunteers will be studied before and after inhalation of wood smoke or clean air for one hour in a purpose built whole-body exposure chamber. The investigators will perform comprehensive vascular assessments thereafter.

Understanding the effects of wood smoke on the blood vessels and clotting will be an important first step in helping to protect firefighters from heart disease. Through research, the investigators hope to identify methods to minimise the risk of heart attacks in firefighters and understand the health effects of a major source of air pollution that is relevant to the general population.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking healthy male firefighters or volunteers

Exclusion Criteria:

* Current smoker or regular users of snus
* History of lung or ischaemic heart disease
* Malignant arrhythmia
* Systolic blood pressure >190mmHg or <100mmHg
* Renal or hepatic dysfunction
* Previous history of blood dyscrasia
* Unable to tolerate the supine position
* Blood donation within the last 3 months
* Recent respiratory tract infection within the past 4 weeks
* Routine medication including aspirin and NSAIDs

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow measured by venous occlusion plethysmography in response to infused vasodilators | 4-6 hours after exposure

SECONDARY OUTCOMES:
Ex-vivo thrombus formation using the Badimon chamber | 2 hours after exposure
Plasma t-PA and PAI concentrations following infusion of bradykinin | During forearm study, 4-6hours after exposure

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas L Mills, MBChB PhD, Study Director — University of Edinburgh; David E Newby, MD PhD, Study Chair — University of Edinburgh; Anders Blomberg, MD PhD, Study Director — Umeå University; Thomas Sandström, MD PhD, Study Director — Umeå Univerisity; Amanda L Hunter, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Umeå University, Umeå, Västerbotten County, Sweden

REFERENCES:
- [Result] Hunter AL, Unosson J, Bosson JA, Langrish JP, Pourazar J, Raftis JB, Miller MR, Lucking AJ, Boman C, Nystrom R, Donaldson K, Flapan AD, Shah AS, Pung L, Sadiktsis I, Masala S, Westerholm R, Sandstrom T, Blomberg A, Newby DE, Mills NL. Effect of wood smoke exposure on vascular function and thrombus formation in healthy fire fighters. Part Fibre Toxicol. 2014 Dec 9;11:62. doi: 10.1186/s12989-014-0062-4. PMID 25487196
- [Derived] Langrish JP, Watts SJ, Hunter AJ, Shah AS, Bosson JA, Unosson J, Barath S, Lundback M, Cassee FR, Donaldson K, Sandstrom T, Blomberg A, Newby DE, Mills NL. Controlled exposures to air pollutants and risk of cardiac arrhythmia. Environ Health Perspect. 2014 Jul;122(7):747-53. doi: 10.1289/ehp.1307337. Epub 2014 Mar 25. PMID 24667535